CLINICAL TRIAL: NCT05820750
Title: Clinical and Radiographic Evaluation of Photodynamic Therapy for Root Canal Treatment of Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Elsayed Abo Farrag, assistant lecturer at paediatric dentistry department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M02041022
Record Dates: First submitted 2023-03-27; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Photodynamic Therapy
MeSH Terms: interventions — Photochemotherapy; Pulpectomy; Metapex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard root canal treatment (Other)
  Interventions: Procedure: pulpectomy with metapex
- photodynamic therapy (Other)
  Interventions: Device: photodynamic therapy
- instrumentation and photodynamic therapy (Other)
  Interventions: Device: photodynamic therapy

INTERVENTIONS:
Device: photodynamic therapy — root canal treatment of primary molars using photodynamic therapy
  Arms: instrumentation and photodynamic therapy; photodynamic therapy
Procedure: pulpectomy with metapex — root canal treatment using standard technique
  Arms: standard root canal treatment

SUMMARY:
This study will be conducted to evaluate clinical and radiographic success of Photodynamic Therapy for root canal treatment of primary molars in comparison to the standard root canal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-7 years.
* Apparent healthy child not suffering from any mental or physical disability.
* Cooperative children.
* Restorable teeth.
* Each child should have at least one carious primary molar with signs and symptoms of irreversible pulpitis or pulp necrosis.
* Absence of internal and / or external perforation in the furcation area.
* At least 2/3 thirds of the roots should be remained.

Exclusion Criteria:

* Children with compromised health or physical disability.
* Resorption of the roots more than 2/3 thirds.
* Non restorable teeth.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical success of photodynamic therapy | 14 months
  The following criteria will be used for the determination of treatment success or failure:
  1. Repair (= success) Clinically: absence of signs and symptoms.
  2. Lack of repair (= failure) Clinically: signs and symptoms indicative of acute apical periodontitis.
Evaluation of radiographic success of photodynamic therapy | 14 months
  The following criteria will be used for the determination of treatment success or failure:
  1. Complete repair (= success) Radiographically: absence of pathological root resorption, normal width of periodontal ligament space, absence of lesion development in periapical regions in cases of absence of lesion in the initial diagnostic radiograph and complete regression of lesion in cases of presence of lesion in the initial diagnostic radiograph.
  2. Incomplete repair (= success) Radiographically: absence of pathological root resorption and reduction lesion size in the periapical region.
  3. Lack of repair (= failure) Radiographically: presence of pathological root resorption, lesion in furcation/periapical region unchanged in size during follow-up period, increase in lesion size or the development of a new lesion.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed El Sayed Abo Farrag, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided